CLINICAL TRIAL: NCT07247058
Title: Isturisa in Management of Mild Autonomous Cortisol Secretion (MACS)
Brief Title: Isturisa Treatment in Mild Autonomous Cortisol Secretion( MACS)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Recordati Rare Diseases Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00511675
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Mild Autonomous Cortisol Secretion (MACS)
Keywords: MACS; Mild Autonomous Cortisol Secretion; Adrenal Adenoma; Osilodrostat; Isturisa; Body Composition; Metabolic Outcomes; Subclinical Cushing Syndrome; Adrenal hyperplasia; Carotid intima thickness; Bone mineral density; Hypertension; Glycemic control
MeSH Terms: conditions — ACTH Syndrome, Ectopic; Adrenal Hyperplasia, Congenital; Hypertension | interventions — Osilodrostat

STUDY DESIGN:
Intervention Model Description: This is a single-arm, interventional study in which all enrolled participants with MACS will receive Osilodrostat (Isturisa). The patients will be evaluated for the impact of Isturisa on clinical features and comorbidities associated with MACS.
Masking Description: This is an open-label study. No parties are masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isturisa Treatment Arm (Experimental): Participants diagnosed with Mild Autonomous Cortisol Secretion (MACS) will receive Osilodrostat (Isturisa) as an investigational treatment. The intervention aims to evaluate comorbidities associated with MACS after the initiation of osilodrostat(Isturisa).
  Interventions: Drug: Osilodrostat (Isturisa)

INTERVENTIONS:
Drug: Osilodrostat (Isturisa) — The intervention aims to evaluate the impact of osilodrostat on cardiometabolic outcomes, bone mineral density, body composition, adrenal tumor size or hyperplasia, and biochemical markers of cortisol excess.
  Other Names: Osilodrostat; Isturisa; LCI699

SUMMARY:
To characterize the impact of Isturisa on clinical features and comorbidities associated with MACS. The investigators hypothesize that patients treated with Isturisa will exhibit significantly better metabolic indicators (such as fasting glucose, HbA1c, and lipid profile), blood pressure, weight, body composition and bone mineral density than at Baseline. The investigators also assess the effect of Isturisa on quality of life and psychological symptoms in patients with MACS. The investigators hypothesize that treatment with Isturisa will lead to significant improvements in quality-of-life scores and reductions in depression scores compared to Baseline.

DETAILED DESCRIPTION:
Mild autonomous cortisol secretion (MACS) is diagnosed in up to 48% of patients with incidentally discovered adrenal tumors or hyperplasia. Based on the finding of adrenal masses in 5% of adults undergoing cross-sectional imaging, the overall prevalence of MACS is about 1-2%. MACS is characterized by autonomous cortisol secretion without the overt symptoms of Cushing syndrome. It is usually associated with low ACTH and DHEAS levels as an indicator of autonomous cortisol secretion. The European Society of Endocrinology-European Network for the Study of Adrenal Tumors (ESE-ENSAT) and the American Association of Clinical Endocrinology (AACE) recommend a cortisol >1.8 μg/dL after 1 mg-DST to define MACS. Several metabolic abnormalities are associated with MACS, including increased cardiovascular disease, mood alteration, hypertension, osteoporosis, hyperglycemia, obesity, weight gain, and lipid abnormalities. Additionally, increased mortality has been reported in MACS patients. Given these complications and increased mortality, there is a need for effective management and treatment options for MACS.

This research aims to evaluate the efficacy and safety of Isturisa in patients with MACS to address the current gap in treatment strategies. By assessing how effectively Isturisa improves cardiometabolic disorders and monitoring its safety profile, the research will seek to provide a clearer understanding of its role as a treatment option in MACS patients who are not a surgical candidate or do not want to pursue surgery. This evaluation is crucial for developing more effective treatment options and improving management strategies for MACS, ultimately contributing to better patient management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years.
* Diagnosis of mild autonomous cortisol secretion (MACS) defined by:
* Serum cortisol >1.8 µg/dL after 1 mg overnight dexamethasone suppression test (DST).
* Presence of adrenal adenoma confirmed by imaging (CT or MRI).
* Ability to provide informed consent.
* Willingness to undergo study procedures including DEXA scan and laboratory assessments.

Exclusion Criteria:

* Known diagnosis of Cushing's syndrome or overt hypercortisolism.
* Current or recent (within 3 months) treatment with glucocorticoids or medications affecting cortisol production (e.g., ketoconazole, metyrapone).
* Severe hepatic impairment or renal failure.
* Pregnancy or breastfeeding.
* Known allergy or contraindication to osilodrostat (Isturisa).
* Participation in another interventional clinical trial within the last 30 days.
* Any medical or psychiatric condition that, in the investigator's judgment, may interfere with study participation or safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in fasting glucose, HbA1c | Baseline, and then every 3 months up to 2 years
  glycemic control: fasting glucose, HbA1c
Change in bone mineral density (g/cm²) | Baseline, 1 year, and 2 years
  Bone mineral density (g/cm²) measured by DEXA scan.
Change in body weight (kg) from baseline during Isturisa treatment | Baseline and every 3 months up to 2 years
  Change in body weight will be measured at baseline and every follow-up visit (approximately every 3 months) throughout the 2-year treatment period with Isturisa.
Change in lipid profile from baseline during Isturisa treatment | Baseline and every 3 months up to 2 years
  Serum lipid profile (LDL-C, HDL-C, total cholesterol, triglycerides) will be assessed at baseline and every follow-up visit (approximately every 3 months) during the 2-year treatment period.
Change in body composition (kg) | baseline, 1 year and 2 years
  Body composition including lean mass and fat mass (kg) measured by DEXA scan.

SECONDARY OUTCOMES:
Change in Quality of Life as assessed by Short Form -36 (SF-36) | Baseline and every 3 months up to 2 years
  Assessment of changes in quality of life using the SF-36 Health Survey. The SF-36 consists of 36 items measuring 8 health domains, with total scores ranging from 0 to 100, where higher scores indicate better quality of life.
Change in carotid intima-media thickness (CIMT) | Baseline, 1 year, and 2 years
  Carotid intima-media thickness (milimeters) will be measured using carotid ultrasound to evaluate vascular changes associated with mild autonomous cortisol secretion. CIMT will be assessed at baseline and at follow-up imaging performed approximately every 12 months during the 2-year treatment period.
Change in adrenal adenoma/hyperplasia size (mm) | Baseline, 1 year, and 2 years
  Adenoma maximal diameter (mm) measured on non-contrast CT at each imaging time point.
Change in Depression Scores as assessed by the Beck Depression Inventory-II | Baseline and every 3 months up to 2 years
  Assessment of changes in depressive symptoms using the Beck Depression Inventory-II (BDI-II). The BDI-II is a 21-item validated questionnaire with total scores ranging from 0 to 63, where higher scores indicate more severe depressive symptoms.

OTHER OUTCOMES:
Change in Inflammatory Biomarkers | Baseline and every 3 months up to 2 years
  Exploratory evaluation of changes in inflammatory biomarkers, specifically high-sensitivity C-reactive protein (hsCRP) and interleukin-6 (IL-6), during treatment with Isturisa in patients with mild autonomous cortisol secretion (MACS). These markers are included in the optional research-specific procedures to assess potential inflammatory or physiologic effects of Isturisa beyond cortisol regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Hamrahian, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feldman D. Ketoconazole and other imidazole derivatives as inhibitors of steroidogenesis. Endocr Rev. 1986 Nov;7(4):409-20. doi: 10.1210/edrv-7-4-409. No abstract available. PMID 3536461
- [Result] Martino M, Aboud N, Lucchetti B, Salvio G, Arnaldi G. Osilodrostat oral tablets for adults with Cushing's disease. Expert Rev Endocrinol Metab. 2022 Mar;17(2):99-109. doi: 10.1080/17446651.2022.2044789. Epub 2022 Feb 28. PMID 35220871
- [Result] Tibblin S, Dymling JF, Ingemansson S, Telenius-Berg M. Unilateral versus bilateral adrenalectomy in multiple endocrine neoplasia IIA. World J Surg. 1983 Mar;7(2):201-8. doi: 10.1007/BF01656143. No abstract available. PMID 6135282
- [Result] Ma L, Yin L, Hu Q. Therapeutic compounds for Cushing's syndrome: a patent review (2012-2016). Expert Opin Ther Pat. 2016 Nov;26(11):1307-1323. doi: 10.1080/13543776.2016.1217331. Epub 2016 Jul 30. PMID 27454103
- [Result] Ren X, Nan M, Zhang X. Evaluating the efficacy of surgical and conservative approaches in mild autonomous cortisol secretion: a meta-analysis. Front Endocrinol (Lausanne). 2024 Jul 17;15:1399311. doi: 10.3389/fendo.2024.1399311. eCollection 2024. PMID 39086899
- [Result] Sbardella E, Minnetti M, D'Aluisio D, Rizza L, Di Giorgio MR, Vinci F, Pofi R, Giannetta E, Venneri MA, Vestri A, Morelli S, Lenzi A, Isidori AM. Cardiovascular features of possible autonomous cortisol secretion in patients with adrenal incidentalomas. Eur J Endocrinol. 2018 May;178(5):501-511. doi: 10.1530/EJE-17-0986. Epub 2018 Mar 6. PMID 29510982
- [Result] Patrova J, Kjellman M, Wahrenberg H, Falhammar H. Increased mortality in patients with adrenal incidentalomas and autonomous cortisol secretion: a 13-year retrospective study from one center. Endocrine. 2017 Nov;58(2):267-275. doi: 10.1007/s12020-017-1400-8. Epub 2017 Sep 8. PMID 28887710
- [Result] Pelsma ICM, Fassnacht M, Tsagarakis S, Terzolo M, Tabarin A, Sahdev A, Newell-Price J, Marina L, Lorenz K, Bancos I, Arlt W, Dekkers OM. Comorbidities in mild autonomous cortisol secretion and the effect of treatment: systematic review and meta-analysis. Eur J Endocrinol. 2023 Oct 17;189(4):S88-S101. doi: 10.1093/ejendo/lvad134. PMID 37801655
- [Result] Czapla-Iskrzycka A, Swiatkowska-Stodulska R, Sworczak K. Comorbidities in Mild Autonomous Cortisol Secretion - A Clinical Review of Literature. Exp Clin Endocrinol Diabetes. 2022 Sep;130(9):567-576. doi: 10.1055/a-1827-4113. Epub 2022 Jul 11. PMID 35817047
- [Result] Vaidya A, Hamrahian A, Bancos I, Fleseriu M, Ghayee HK. THE EVALUATION OF INCIDENTALLY DISCOVERED ADRENAL MASSES. Endocr Pract. 2019 Feb;25(2):178-192. doi: 10.4158/DSCR-2018-0565. PMID 30817193
- [Result] Fassnacht M, Tsagarakis S, Terzolo M, Tabarin A, Sahdev A, Newell-Price J, Pelsma I, Marina L, Lorenz K, Bancos I, Arlt W, Dekkers OM. European Society of Endocrinology clinical practice guidelines on the management of adrenal incidentalomas, in collaboration with the European Network for the Study of Adrenal Tumors. Eur J Endocrinol. 2023 Jul 20;189(1):G1-G42. doi: 10.1093/ejendo/lvad066. PMID 37318239
- [Result] Trandafir AI, Ghemigian A, Ciobica ML, Nistor C, Gurzun MM, Nistor TVI, Petrova E, Carsote M. Diabetes Mellitus in Non-Functioning Adrenal Incidentalomas: Analysis of the Mild Autonomous Cortisol Secretion (MACS) Impact on Glucose Profile. Biomedicines. 2024 Jul 18;12(7):1606. doi: 10.3390/biomedicines12071606. PMID 39062179
- [Result] Zavatta G, Vicennati V, Altieri P, Tucci L, Colombin G, Coscia K, Mosconi C, Balacchi C, Fanelli F, Malagrino M, Magagnoli M, Golfieri R, Pagotto U, Di Dalmazi G. Mild autonomous cortisol secretion in adrenal incidentalomas and risk of fragility fractures: a large cross-sectional study. Eur J Endocrinol. 2023 Apr 4;188(4):343-352. doi: 10.1093/ejendo/lvad038. PMID 36952249
- [Result] Delivanis DA, Athimulam S, Bancos I. Modern Management of Mild Autonomous Cortisol Secretion. Clin Pharmacol Ther. 2019 Dec;106(6):1209-1221. doi: 10.1002/cpt.1551. Epub 2019 Aug 6. PMID 31206616